CLINICAL TRIAL: NCT07005232
Title: Lead Evaluation for Defibrillation and Reliability Post Approval Study (LEADR PAS)
Brief Title: Lead Evaluation for Defibrillation and Reliability Post Approval Study
Acronym: LEADR PAS
Status: Enrolling by invitation | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: LEADR PAS
Record Dates: First submitted 2025-05-21; First posted 2025-06-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-05

CONDITIONS: Tachyarrhythmia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: defibrillation lead — This is a device registry for the OmniaSecure™ defibrillation lead. The OmniaSecure lead is a steroid eluting, integrated bipolar, nonretractable screw-in, catheter delivered, transvenous ventricular lead with a Right Ventricular (RV) defibrillation coil electrode. The lead is designed for pacing, sensing, cardioversion, and defibrillation therapies, and has application for patients whom transvenous ICDs and cardiac resynchronization therapy defibrillators (CRT-Ds) are indicated.

SUMMARY:
Medtronic is sponsoring the LEADR PAS to provide continuing evaluation and periodic reporting of safety and effectiveness of the OmniaSecure™ defibrillation lead following commercial release. The LEADR PAS is conducted within Medtronic's Product Surveillance Registry Platform (NCT01524276).

DETAILED DESCRIPTION:
The LEADR PAS is a global, prospective, observational, multi-site registry study. This study is conducted within Medtronic's Product Surveillance Registry Platform (NCT01524276).

Eligibility for enrollment is based on market release dates for the OmniaSecure™ defibrillation lead within the geography in which the subject is enrolled.

Patients enrolled in LEADR PAS will be prospectively followed for the lifetime of device post-implant or until registry closure, patient death, or patient exit from the registry (i.e., withdrawal of consent).

Successfully implanted patients are expected to have scheduled follow-up visits per routine clinical care, at least annually, or as prompted by reportable adverse events. The primary objective analysis will occur when 500 patients reach 5 years of follow-up. The total estimated registry duration is through lifetime of device.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has, or is intended to receive or be treated with an OmniaSecure™ defibrillation lead.
* Patient is consented prior to or within 30 days of the therapy received or consented as continuation from the LEADR Pivotal study

Exclusion Criteria:

* Patient who is, or is expected to be, inaccessible for follow-up
* Patient is excluded by local local law
* Patient is currently enrolled or plans to enroll in any concurrent drug and/or device study that may confound the Product Surveillence Registyr (PSR) results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Geographies with regulatory approval for the OmniaSecure™ defibrillation lead are eligible to enroll patients (see locations section). Any patient receiving an implant of the OmniaSecure lead, based on the treating physician's medical discretion, is eligible for enrollment into the study (patients previously enrolled in the pre-market clinical trial with a clinical model 093000 OmniaSecure lead may also be eligible for continued follow-up into the OmniaSecure PAS). In geographies where applicable, OmniaSecure PAS will include adolescent pediatric patients, who are at least 30 kg and are also at least 12 years of age, whose cardiac anatomy is conducive to RV coil placement.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2032-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Complication Survival Rate | 5 years
  Estimate OmniaSecure lead-related complication-free survival through 5 years post implant.

CONTACTS AND LOCATIONS:
Locations (29):
- United States (28):
  - COR Healthcare, Torrance, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Hartford Hosptial, Hartford, Connecticut
  - University of South Florida Health (USF), Tampa, Florida
  - Iowa Heart Center (West Des Moines IA), West Des Moines, Iowa
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Metropolitan Cardiology Consultants, Coon Rapids, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - North Memorial Health Heart & Vascular Center, Robbinsdale, Minnesota
  - Saint Lukes Health System, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Virtua Health, Marlton, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - Northwell Health South Shore University Hospital, Bay Shore, New York
  - Northwell Health Huntington Hospital, Huntington, New York
  - Northwell Health Staten Island University Hospital, Staten Island, New York
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
- Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No